CLINICAL TRIAL: NCT03628911
Title: Evaluation of the Ongoing Safety and Preliminary Efficacy of the Tetanizing Burst Therapy (TBT) System in Subjects Undergoing ICD Replacement Due to End-of-battery Life
Brief Title: Study to Evaluate Tetanizing Burst Therapy in Patients Undergoing ICD Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EP Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBT001
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Electrophysiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Tetanizing Burst Therapy — Tetanizing Burst Therapy tetanizes skeletal muscle with a brief burst of stimulation prior to ICD shock, thereby reducing muscular contraction due to the shock

SUMMARY:
This study evaluates whether the addition of tetanizing burst therapy reduces the pain associated with ICD shocks

DETAILED DESCRIPTION:
The implantable cardioverter defibrillator is a device designed to rescue patients from life-threatening arrhythmias by delivering a defibrillation shock to allow restoration of cardiac rhythm. These defibrillation shocks are extremely painful, owing to sudden rapid contraction of thoracic and abdominal skeletal muscle, which, in addition to the heart, are stimulated by the defibrillation shock. Tetanizing Burst Therapy is a novel electrical waveform which tetanizes skeletal muscle with a brief burst of stimulation prior to the ICD shock, thereby reducing muscular contraction due to the shock. This study is designed for those patients who are already undergoing ICD replacement.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18-80 years, inclusive
* Ability to understand and provide written informed consent
* Normal sinus rhythm
* Standard transvenous left-sided ICD referred for device replacement due to end of battery life

Exclusion Criteria:

* Heart rate <40 or >90 bpm
* Atrial fibrillation or pacemaker dependent
* NYHA Class III/IV symptoms of HF
* MI within 90 days of enrollment
* Severe cardiac ischemia manifested by chest pain at rest or with minimal exercise
* History stroke or TIAs
* History of prior ICD pocket infection
* ICD lead resistance that is too high or too low in the opinion of the investigator
* Female who is pregnant or breastfeeding
* Prior heart transplant
* Serum electrolytes out of normal range at participating institution

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Less pain after TBT impulse with ICD shock compared to ICD shock alone | 5 minutes
  Each subject will receive 2 therapies in random order delivered 5 minutes apart:
  * Tetanizing Burst Therapy + shock; and
  * Pure shock alone. Using the Numeric Pain Rating Scale (NRS) after each shock, the subject will be asked to provide a verbal score between 1 and 10, where 1 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
The efficacy of tetanizing burst therapy in subjects undergoing ICD replacement as assessed by NRS verbal score | 5 minutes
  After each shock, a blinded assessor will ask the subject to provide an NRS verbal score between 1 and 10, where 1 is no pain and 10 is the worst pain imaginable. The percent change in the NRS score will be calculated for each subject along with the change in skeletal muscle force waveform
The safety of tetanizing burst therapy in subjects undergoing ICD replacement as assessed by adverse events | 7 days
  Incidence rates of all adverse events will be calculated and compared to event rates in the literature. They will also be analyzed by severity and relationship to the device and/or study procedures.
The device performance of tetanizing burst therapy in subjects undergoing ICD replacement as assessed degree of muscle contraction (Rate of Force Development) | 5 minutes
  The force of contraction is recorded at the patient's left elbow with a myometer

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Berger, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No